CLINICAL TRIAL: NCT02072668
Title: The Effect of Factor Xa Inhibition, With Rivaroxaban, on the Pathology of Sickle Cell Disease
Brief Title: The Effect of Rivaroxaban in Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-2607; U01HL117659-01 (NIH)
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Sickle Cell Anemia; Sickle Cell-Beta0-Thalassemia
Keywords: sickle cell anemia; sickle cell disease; rivaroxaban; direct Xa inhibition; coagulation; anticoagulation
MeSH Terms: conditions — Anemia, Sickle Cell; Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban for 4 wks, Placebo for 4 wks (Other): Subject will receive rivaroxaban 20mg PO daily for 4 weeks and then matching placebo 1 PO daily for 4 weeks, with a 2-week wash out period in between the two treatment phases. Both of the two treatments will be in capsule form.
  Interventions: Drug: rivaroxaban; Drug: placebo
- Placebo for 4 wks, rivaroxaban for 4 wks (Other): Subject will receive placebo 1 PO daily for 4 weeks, then rivaroxaban 20mg PO daily for 4 weeks, with a 2-week wash out period in between the two treatment phases. Both of the two treatments will be in capsule form.
  Interventions: Drug: rivaroxaban; Drug: placebo

INTERVENTIONS:
Drug: rivaroxaban — Subject will receive rivaroxaban 20mg PO daily for 4 weeks and then matching placebo 1 PO daily for 4 weeks, with a 2-week wash out period in between the two treatment phases. Both of the two treatments will be in capsule form OR Subject will receive placebo 1 PO daily for 4 weeks, then rivaroxaban 20mg PO daily for 4 weeks, with a 2-week wash out period in between the two treatment phases. Both of the two treatments will be in capsule form.
  Other Names: Xarelto
Drug: placebo — Subject will receive rivaroxaban 20mg PO daily for 4 weeks and then matching placebo 1 PO daily for 4 weeks, with a 2-week wash out period in between the two treatment phases. Both of the two treatments will be in capsule form OR Subject will receive placebo 1 PO daily for 4 weeks, then rivaroxaban 20mg PO daily for 4 weeks, with a 2-week wash out period in between the two treatment phases. Both of the two treatments will be in capsule form.

SUMMARY:
The primary study hypothesis is that inhibition of factor Xa with rivaroxaban will reduce inflammation, coagulation and endothelial cell activation, and improve microvascular blood flow in patients with sickle cell disease (SCD) during the non-crisis, steady state. To test this hypothesis, this study will evaluate the effects of rivaroxaban on:

* plasma markers of inflammation;
* plasma markers of endothelial activation;
* plasma markers of thrombin generation; and
* microvascular blood flow assessed using laser Doppler velocimetry (LDV) of post-occlusive reactive hyperemia (PORH).

In a cross-over design, subjects will receive rivaroxaban 20 mg/day and placebo for 4 weeks each, separated by a 2-week washout phase.

DETAILED DESCRIPTION:
The study will consist of a Screening Phase, two Treatment Phases, a Wash-Out Phase, and a Follow-up Phase. The Screening Phase will occur within 28 days of randomization and will include informed consent, a physical examination, and complete medical history to include determination of sickle cell genotype and current medications. Clinical laboratory tests to be performed include: a Complete Blood Count (CBC) with differential and reticulocyte count; Prothrombin time(PT) / activated partial thromboplastin time (aPTT); and serum chemistries (BUN, creatinine, total and direct bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and LDH). A chest x-ray and MRI/MRA of the brain will also be done at Screening to rule out underlying disease.

If the patient is found through the screening process to be eligible, the 1st Treatment Phase begins. Baseline safety assessments and measurement of biomarkers are completed, then the subject is randomized to receive rivaroxaban or placebo. After 4 weeks of treatment, there is a 2-Week Wash-Out Phase. After the Wash-Out Phase, another set of baseline studies are performed and the 2nd Treatment Phase begins. For this Phase of the study, the subject "crosses over" to receive whatever treatment - rivaroxaban or placebo - that they did not receive in the 1st Treatment Phase. After taking the assigned study drug for 4 weeks, the 2nd Treatment Phase ends. The subject returns 2 weeks after the last dose of study treatment for the Follow-Up Phase, consisting of a single end-of-study visit during which safety assessments are repeated.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age; sickle cell anemia (HbSS) or sickle-beta0 (HbSβ0) thalassemia;
* serum creatinine ≤ 1.0 mg/dL men) or 1.2 mg/dL (women);
* ALT </= 2 times upper limits of normal;
* platelet count ≥ 50,000 cu/mm;
* normal baseline PT/international normalized ratio (INR) and aPTT;
* be in the non-crisis, "steady state" with no severe pain episodes during the preceding 4 weeks;
* ability to understand the requirements of the study and be willing to give informed consent;
* women of childbearing age must be practicing an adequate method of contraception;
* and if on hydroxyurea, be on a stable dose for at least 3 months prior to enrollment.

Exclusion Criteria:

* hypersensitivity to any component of rivaroxaban;
* history of major GI bleeding or bleeding diathesis;
* baseline Hb < 5.5 gm/dL;
* history of clinically overt stroke;
* brain magnetic resonance imaging with angiography (MRI/MRA) scan with evidence of Moya Moya;
* pregnant or breastfeeding;
* active liver disease or ALT > 3 times upper limit of normal;
* on chronic anticoagulant, non-steroidal anti-inflammatory (NSAID) or statin therapy;
* history of metastatic cancer;
* current alcohol abuse;
* on a chronic transfusion program or any blood transfusion in the 3 months prior to enrollment;
* ingested any investigational drugs within the past 4 weeks;
* use of CYP3A4/P-glycoprotein inducers such as carbamazepine, phenytoin, rifampin, and St John's wort;
* use of CYP3A4/P- glycoprotein inhibitors such as ketoconazole, indinavir/ritonavir, itraconazole, lopinavir/ritonavir, ritonavir, and conivaptan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-02; Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth I Ataga, MBBS, Principal Investigator — University of North Carolina, Chapel Hill; Nigel Key, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Ataga KI, Elsherif L, Wichlan D, Wogu AF, Matsui N, Pawlinski R, Cai J, Key NS. A pilot study of the effect of rivaroxaban in sickle cell anemia. Transfusion. 2021 Jun;61(6):1694-1698. doi: 10.1111/trf.16343. Epub 2021 Mar 4. PMID 33660875

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 subjects signed informed consent and were successfully screened. One subject withdrew during Baseline and prior to the first intervention and data from this individual are included in the baseline characteristics. One subject entered the second intervention period but was lost to follow up before receiving the intervention.
Groups:
- Rivaroxaban, Then Placebo: Participants first received Rivaroxaban 20 mg tablet once daily for 4 weeks. After a washout period of 2 weeks, they then received placebo (matching Rivaroxaban 20 mg tablet) once daily for 4 weeks.
  Rivaroxaban: 20 mg tablet by mouth daily for 4 weeks Placebo: Matching placebo tablet by mouth daily for 4 weeks
- Placebo, Then Rivaroxaban: Participants first received placebo (matching Rivaroxaban 20 mg tablet) once daily for 4 weeks. After a washout period of 2 weeks, they then received Rivaroxaban 20 mg tablet once daily for 4 weeks.
  Rivaroxaban: 20 mg tablet by mouth daily for 4 weeks Placebo: Matching placebo tablet by mouth daily for 4 weeks
Period: First Intervention
Arm/Group | Rivaroxaban, Then Placebo | Placebo, Then Rivaroxaban
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Rivaroxaban, Then Placebo | Placebo, Then Rivaroxaban
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Rivaroxaban, Then Placebo | Placebo, Then Rivaroxaban
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who had a screening visit
Groups:
- Study Participants: Participants who had a screening visit
Arm/Group | Study Participants
Number analyzed (Participants) | 15
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 39.00 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 68.22 (11.69)
Height [Mean (Standard Deviation); unit: cm] — Population: Only measured on the participants who received study medication
  cm
    number analyzed (Participants) | 14
    (all) | 169.40 (10.56)
White Blood Cell (WBC) count [Mean (Standard Deviation); unit: 10^9 cells/L] | 8.49 (2.03)
Genotype - Hemoglobin SS (HbSS) [Count of Participants; unit: Participants] | 15
Platelet count [Mean (Standard Deviation); unit: 10^9 cells/L] | 370.07 (169.13)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.22)
Prothrombin Time (PT) [Mean (Standard Deviation); unit: sec] — A test that measures how quickly blood clots Population: Only measured on the participants who received study medication
  sec
    number analyzed (Participants) | 14
    (all) | 12.54 (0.99)
International Normalized Ratio (INR) [Mean (Standard Deviation); unit: ratio] — The ratio of a patient's prothrombin time to a normal (control) sample Population: Only measured on the participants who received study medication
  ratio
    number analyzed (Participants) | 14
    (all) | 1.13 (0.09)
Partial Thromboplastin Time (PTT) [Mean (Standard Deviation); unit: sec] — Measures the time it takes for a blood clot to form Population: Only measured on the participants who received study medication
  sec
    number analyzed (Participants) | 14
    (all) | 27.16 (2.48)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Weeks in Soluble Vascular Cell Adhesion Molecule-1 (VCAM-1)
Description: Assay performed for soluble VCAM-1 using a commercially available enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline, 4 weeks
Population: Data reported only for those participants who completed both interventions.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Rivaroxaban: Participants who received Rivaroxaban 20 mg tablet in either the first or the second half of the study
- Placebo: Participants who received placebo tablet (matching Rivaroxaban 20 mg) in either the first or the second half of the study
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 13 | 13
pg/mL | 40.9 [-115.5 to 197.2] | 10.7 [-84.5 to 105.8]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.6281, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

2. Primary Outcome: Change From Baseline to 4 Weeks in Interleukin-6 (IL-6)
Description: Assay performed for IL-6 using a commercially available enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline, 4 weeks
Population: Data reported only for those participants who completed both interventions.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 13 | 13
pg/mL | -1.1 [-4.47 to 2.28] | -0.54 [-1.69 to 0.62]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.7973, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

3. Secondary Outcome: Change From Baseline to Week 4 in the Plasma Marker of Inflammation IL-2
Description: Interleukin-2 (IL-2) was measured using Luminex MAP technology at the UNC core facility
Time Frame: Baseline, 4 weeks
Population: Data analyzed for the 13 participants completing both interventions but results for 6 participants in each group fell outside the standard curve and could not be extrapolated.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 7 | 7
pg/mL | -1.14 [-4.13 to 1.85] | 0.36 [-3.48 to 4.2]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.4442, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

4. Secondary Outcome: Change From Baseline to Week 4 in the Plasma Marker of Inflammation IL-8
Description: Interleukin-8 (IL-8) was measured using Luminex MAP technology at the UNC core facility
Time Frame: Baseline, 4 weeks
Population: Data analyzed for the 13 participants completing both interventions but results for 4 participants in the rivaroxaban group and 5 participants in the placebo group fell outside the standard curve and could not be extrapolated.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 9 | 8
pg/mL | 0.95 [-41.83 to 43.72] | -4.08 [-38.36 to 30.19]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.2545, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

5. Secondary Outcome: Change From Baseline to Week 4 in Plasma Marker of Inflammation hsCRP
Description: high sensitivity C-reactive protein (hsCRP) was measured using Luminex MAP technology at the UNC core facility.
Time Frame: Baseline, 4 weeks
Population: Biomarker evaluations were limited to IL-2 and IL-8 as those were thought more likely to reflect inflammation activation based on experience in recent studies.
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline to Week 4 in Plasma Marker of Inflammation MPO
Description: myeloperoxidase (MPO) was measured using Luminex MAP technology at the UNC core facility.
Time Frame: Baseline, 4 weeks
Population: as for outcome 5
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline to Week 4 in Plasma Marker of Inflammation TNF-a
Description: tumor necrosis factor alpha (TNF-a) was measured using Luminex MAP technology at the UNC core facility.
Time Frame: Baseline, 4 weeks
Population: as for outcome 5
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline to Week 4 in Plasma Marker of Inflammation sPLA2
Description: secretory phospholipase A2 (sPLA2) was measured using Luminex MAP technology at the UNC core facility
Time Frame: Baseline, 4 weeks
Population: as for outcome 5
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline to Week 4 in Marker of Endothelial Cell (EC) Activation sICAM
Description: levels of soluble intracellular adhesion molecule (sICAM) were measured using a commercially available ELISA
Time Frame: Baseline, 4 weeks
Population: Biomarker evaluations were limited to VCAM-1 and IL-6 as those were thought more likely to reflect endothelial cell activation based on experience in recent studies.
Arm/Group | Rivaroxaban, Then Placebo | Placebo, Then Rivaroxaban
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline to Week 4 in TH1
Description: Microvascular blood flow was measured using laser doppler velocimetry (LDV) assessments of post-occlusive reactive hyperemia (PORH). This was accomplished using the Perimed PF5001 Velocitometer (Stockholm, Sweden). Variable measured: time to half before hyperemia (TH1)
Time Frame: Baseline, 4 weeks
Population: All participants randomized to each treatment were analyzed.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 14 | 13
seconds | 0.84 [-0.79 to 2.47] | -0.51 [-2.72 to 1.7]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.4374, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

11. Secondary Outcome: Change From Baseline to Week 4 in TM
Description: Microvascular blood flow was measured using laser doppler velocimetry (LDV) assessments of post-occlusive reactive hyperemia (PORH). This was accomplished using the Perimed PF5001 Velocitometer (Stockholm, Sweden). Variable measured: time to max (TM)
Time Frame: Baseline, 4 weeks
Population: All participants randomized to each treatment were analyzed.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 14 | 13
seconds | -0.97 [-5.71 to 3.77] | -2.01 [-6.82 to 2.81]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.3470, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

12. Secondary Outcome: Change From Baseline to Week 4 in AH
Description: Microvascular blood flow was measured using laser doppler velocimetry (LDV) assessments of post-occlusive reactive hyperemia (PORH). This was accomplished using the Perimed PF5001 Velocitometer (Stockholm, Sweden). Variable measured: hyperemia area (AH)
Time Frame: Baseline, 4 weeks
Population: All participants randomized to each treatment were analyzed.
Measure: Mean (95% Confidence Interval); unit: perfusion units*seconds
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 14 | 13
perfusion units*seconds | 128 [-373 to 628] | -1189 [-2597 to 218]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.0755, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

13. Secondary Outcome: Change in Ratio From Baseline to Week 4 in AH/AO
Description: Microvascular blood flow was measured using laser doppler velocimetry (LDV) assessments of post-occlusive reactive hyperemia (PORH). This was accomplished using the Perimed PF5001 Velocitometer (Stockholm, Sweden). Variables measured: hyperemia area (AH) and occlusion area (AO)
Time Frame: Baseline, 4 weeks
Population: All participants randomized to each treatment were analyzed.
Measure: Mean (95% Confidence Interval); unit: ratio of AH to AO
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 14 | 13
ratio of AH to AO | 0.05 [-0.46 to 0.57] | -0.81 [-2.05 to 0.42]

14. Secondary Outcome: Change From Baseline to Week 4 in PF
Description: Microvascular blood flow was measured using laser doppler velocimetry (LDV) assessments of post-occlusive reactive hyperemia (PORH). This was accomplished using the Perimed PF5001 Velocitometer (Stockholm, Sweden). Variable measured: peak flow (PF)
Time Frame: Baseline, 4 weeks
Population: All participants randomized to each treatment were analyzed.
Measure: Mean (95% Confidence Interval); unit: perfusion units
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 14 | 13
perfusion units | 3.14 [-9.08 to 15.36] | -12.62 [-26.63 to 1.4]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.0708, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

15. Secondary Outcome: Change From Baseline to Week 4 in RF
Description: Microvascular blood flow was measured using laser doppler velocimetry (LDV) assessments of post-occlusive reactive hyperemia (PORH). This was accomplished using the Perimed PF5001 Velocitometer (Stockholm, Sweden). Variable measured: rest flow (RF)
Time Frame: Baseline, 4 weeks
Population: All participants randomized to each treatment were analyzed.
Measure: Mean (95% Confidence Interval); unit: perfusion units
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 14 | 13
perfusion units | 0.29 [-1.47 to 2.05] | -0.62 [-2.96 to 1.73]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.4501, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

16. Secondary Outcome: Change From Baseline to Week 4 in TAT
Description: Assay for thrombin antithrombin (TAT) complexes performed using commercially available enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline, 4 weeks
Population: Data reported only for those participants who completed both interventions.
Measure: Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 13 | 13
ug/mL | -34.44 [-69.4 to 0.53] | 0.35 [-3.77 to 4.47]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.0767, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

17. Secondary Outcome: Change From Baseline to Week 4 in D-Dimer
Description: Assay for D--dimer is performed using commercially available enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline, 4 weeks
Population: Data reported only for those participants who completed both interventions.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 13 | 13
ng/mL | -471 [-1654 to 712] | -1035 [-3880 to 1810]
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Test type: Superiority; p = 0.7250, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

ADVERSE EVENTS:
Time Frame: Data collected from date of informed consent to end of study visit, approximately 3 months
Description: The safety analysis population includes all participants exposed to any study intervention evaluated in this study.
Arm/Group | Rivaroxaban | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/13
Other Adverse Events (participants affected / at risk) | 8/14 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (N=14) | Placebo (N=13)
painful crisis with bacteremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (N=14) | Placebo (N=13)
pain crisis treated at home (Vascular disorders) | 4 (6) | 2 (2)
headache (General disorders) | 2 (2) | 1 (1)
chest pain (General disorders) | 3 (3) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
ankle laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
tick bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
diarrhea, nausea and vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
insomnia (General disorders) | 1 (1) | 0 (0)
tinea versicolor (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
elevate liver enzymes (Gastrointestinal disorders) | 0 (0) | 1 (1)
cough, fever, body aches, congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
pain in lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
dyspnea (General disorders) | 1 (1) | 0 (0)
pelvic pressure with urination (Renal and urinary disorders) | 1 (1) | 0 (0)
right flank pain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT02072668/Prot_SAP_000.pdf